CLINICAL TRIAL: NCT01808014
Title: The Analgesic Effect of Nefopam on the Fentanyl Based PCA (Patient-controlled Analgesia) After Lumbar Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2012-0920
Record Dates: First submitted 2013-02-27; First posted 2013-03-08 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Lumbar Spinal Stenisis or Lumbar Herniated Intervertebral Disc
Keywords: nefopam, spinal surgery, postoperative pain control
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The addition of Nefopam (Experimental): The addition of Nefopam for intravenous patient-controlled analgesia in patients with lumbar spinal surgery would reduce the side effects seen in monotherapy with opioid analgesia and result in effective pain management.
  Interventions: Drug: nefopam

INTERVENTIONS:
Drug: nefopam — The chief investigator prepared the medications according to the selected randomized table, and investigators who were not involved in medication preparation recorded the pain and prevalence of complications in study subjects. The double-blind restriction was lifted if the patient withdrew from the study, and the next patient was classified into a group while blinded by using the randomized table.Intramuscular midazolam 0.05 mg/kg was administered as a premedication, and then a blood pressure machine, electrocardiogram, and pulse oximeter were connected to the patient in the operating room.

SUMMARY:
Posterior lumbar spinal surgical pain leads to a severe degree of pain, and, hence, various means of pain management are required. Opioid pain medications such as morphine and fentanyl are frequently used as intravenously administered medications. To reduce the use of opioids for pain relief, a non-opioid form of pain relief, such as a Non-Steroidal Anti-Inflammatory Drug (NSAID), is often added to the regimen.

With the use of NSAIDs, however, the risk of systemic side effects such as bleeding, gastroduodenal bleeding, and kidney damage are being reported, and there is also a report of inhibition of spinal fusion; these risks limit the use of NSAIDs.

Nefopam, a new centrally-acting analgesic agent, has been reported in an animal study to desensitize post-surgical pain, and when used with an opioid analgesic, it indirectly controlled the NMDA receptor, which inhibited the generation of c-fos gene at the spine. There are also reports that Nefopam managed pain by inhibiting the serotonin reuptake receptors.

In clinical practice, the administration of Nefopam in patients who required post-surgical pain management reduced the use of opioid analgesics by 20-50 % and also reduced the prevalence of nausea and vomiting.

Therefore, the investigators considered whether the addition of Nefopam for intravenous patient-controlled analgesia in patients with lumbar spinal surgery would reduce the side effects seen in monotherapy with opioid analgesia and result in effective pain management. This study was conducted to address this question.

ELIGIBILITY:
A. Inclusion criteria: The study subjects were adult patients, 20-65 years old, who were going to have spinal fusion surgery due to conditions such as spinal stenosis or disks and who fell under the American Society of Anesthesiologist physical status classifications of 1 or 2.

B. Exclusion criteria: Patients who could not read or understand the consent documents or who had a defect in blood coagulation, hepatectomy, pneumonectomy, nephrectomy, cardiovascular disease, administration of MAO inhibitor, ischuria, glaucoma, or a history of seizure were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The additional analgesic effect of nefopam on the fentanyl based PCA after lumbar spinal surgery | up to 48 hours post-surgery
  The resting visual analogue scale (r-VAS) and cough visual analogue scale (c-VAS) were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea